CLINICAL TRIAL: NCT02341560
Title: A Phase 2/3, Randomized, Double-Masked, Sham-Controlled Trial of QPI-1007 Delivered By Single or Multi-Dose Intravitreal Injection(s) to Subjects With Acute Nonarteritic Anterior Ischemic Optic Neuropathy (NAION)
Brief Title: Phase 2/3, Randomized, Double-Masked, Sham-Controlled Trial of QPI-1007 in Subjects With Acute Nonarteritic Anterior Ischemic Optic Neuropathy (NAION)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: An interim analysis did not warrant to continue enrollment
Sponsor: Quark Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QRK207
Record Dates: First submitted 2015-01-13; First posted 2015-01-19 (Estimated); Last update posted 2020-07-20 (Actual); Status verified 2019-07

CONDITIONS: Non Arteritic Anterior Ischemic Optic Neuropathy
Keywords: NAION
MeSH Terms: conditions — Optic Neuropathy, Ischemic | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- single dose or multiple dose (Active Comparator): QPI-1007 Injection - 1.5 mg
  Interventions: Drug: QPI-1007 Injection - 1.5 mg
- single or multiple dose (Active Comparator): QPI-1007 Injection - 3.0 mg
  Interventions: Drug: QPI-1007 Injection - 3.0 mg
- Sham (Sham Comparator): Sham injection procedure
  Interventions: Other: Sham Injection Procedure

INTERVENTIONS:
Drug: QPI-1007 Injection - 1.5 mg
  Other Names: QPI-1007
  Arms: single dose or multiple dose
Drug: QPI-1007 Injection - 3.0 mg
  Other Names: QPI-1007
  Arms: single or multiple dose
Other: Sham Injection Procedure — Sham Procedure
  Other Names: Sham
  Arms: Sham

SUMMARY:
This study will determine the effect of QPI-1007 on visual function in subjects with recent-onset NAION and assess the safety and tolerability of intravitreal injections of QPI-1007 in this population. This study will also evaluate the structural changes in the retina following administration of QPI-1007.

DETAILED DESCRIPTION:
This is a double masked, randomized, sham-controlled efficacy and safety study that will enroll approximately 800 subjects with recent-onset NAION. Subjects will be randomized into one of 3 groups in a 1:1:1 ratio, and assigned to receive QPI-1007 and/or a sham procedure. Subjects will have a two in three (66%) chance of receiving active treatment (no sham procedure) and a one in three (33%) chance of receiving sham procedure (no active treatment). Total study time involvement is approximately 12 months.

ELIGIBILITY:
Key Inclusion Criteria:

* Positive diagnosis of first episode of NAION in the study eye with symptom onset within 14 days prior to planned study drug administration/sham procedure
* Best corrected visual acuity score in the study eye is better than or equal to 15 letter score, measured using the ETDRS visual acuity protocol at Day 1 prior to study drug administration/sham procedure.
* Clear ocular media and able to undergo adequate pupil dilation to allow a good fundus examination

Key Exclusion Criteria:

* Present use or history of any treatment for the current episode of NAION, including systemic steroids, brimonidine, or traditional Chinese herbal medicine
* Prior episode of NAION in the study eye only
* Present use of drugs known to cause optic nerve or retinal toxicity at Day 1/Randomization, such as: chloroquine or hydroxychloroquine, ethambutol, Vigabatrin. Subjects who need to be prescribed any of these drugs during the course of the study will be discontinued from the trial.
* Any medical condition, concomitant therapy, or previous incisional or laser surgery that, in the opinion of the Investigator, would preclude IVT injection in the study eye only
* Clinical evidence of temporal arteritis

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 732 (Actual)
Dates: Start 2016-02-24 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Effect of QPI-1007 as assessed by Best Corrected Visual Acuity (BCVA) | Baseline through Month 12
Safety and tolerability of QPI-1007 as assessed by adverse events (AE), laboratory evaluations, ECGs, ophthalmic evaluations, slit lamp anterior/posterior examinations, intraocular pressure measurements, presence/absence of vitreous inflammation | Baseline through Month 12

SECONDARY OUTCOMES:
Mean change in BCVA score, as measured by ETDRS visual acuity protocol in the study eye | Day 1 through Month 12
Mean change of Visual Fields, as assessed by Humphrey standard automated perimetry | Day 1 through Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Klier, M.D., Study Director — Quark Pharmaceuticals
Locations (85):
- United States (44):
  - University of Arkansas Medical Center, Jones Eye Institute, Little Rock, Arkansas
  - Loma Linda University Eye Institute, Loma Linda, California
  - University of Southern California, Los Angeles, California
  - NeuroEyeOrbit Institute, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Unversity of California, Los Angeles (UCLA), Pasadena, California
  - University of Colorado Denver, Department of Neurology, Aurora, Colorado
  - Retina Consultants of Southern Colorado, PC, Colorado Springs, Colorado
  - The Eye Care Group, Waterbury, Connecticut
  - Cape Coral Eye Center, Cape Coral, Florida
  - University of Miami Miller School of Medicine/Bascom Palmer Eye Institute, Miami, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Northwestern University, Chicago, Illinois
  - University of Illinois at Chicago, Department of Ophthalmology (MC 648), Chicago, Illinois
  - NorthShore University Healthsystem, Glenview, Illinois
  - University of Kentucky, Department of Neurology, Lexington, Kentucky
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Bethesda Neurology, LLC, Bethesda, Maryland
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - University of Nebraska Medical Center and Truhlsen Eye Institute, Omaha, Nebraska
  - Rutgers, New Jersey Medical School, Newark, New Jersey
  - New York Eye and Ear Infirmary of Mount Sinai, New York, New York
  - Cornell University School of Medicine, New York, New York
  - University of Rochester, Flaum Eye Institute, Rochester, New York
  - State University of New York at Stony Brook, Stony Brook, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Duke University Eye Center, Durham, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Cleveland Clinic, Cole Eye Institute, Cleveland, Ohio
  - Dean McGee Eye Institute, Oklahoma City, Oklahoma
  - University of Pennsylvania, Scheie Eye Institute, Philadelphia, Pennsylvania
  - Retina Consultants of Charleston, Charleston, South Carolina
  - University of Houston, Neuro-Ophth of Texas, Houston, Texas
  - Houston Methodist Hospital, Blanton Eye Institute, Houston, Texas
  - Foresight Studies, San Antonio, Texas
  - University of Utah John A. Moran Eye Center, Salt Lake City, Utah
  - University of Virginia Health Sciences Center, Charlottesville, Virginia
  - Swedish Medical Center, CO/NOCNW, Seattle, Washington
  - University of Washington Department of Ophthalmology, Seattle, Washington
- Australia (4):
  - Sydney Eye Hospital/Save Sight Institute, Sydney, New South Wales
  - Vision South Australia, Kent Town, South Australia
  - The Royal Victorian Eye and Ear Hospital, Fitzroy, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- China (5):
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Peking University Eye Center, The Third Hospital Peking University., Beijing
  - Beijing Tongren Hospital, Capital Medical University, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Tianjin Eye Hospital, Tianjin
- Germany (6):
  - Universitätsmedizin d. Johannes Gutenberg-Universität Mainz, Mainz, Rhineland-Palatinate
  - Universitätsklinikum Aachen-Augenklinik, Aachen
  - Universitätsklinikum Carl Gustav Carus-Dresden-Klinik und Poliklinik für Augenheilkunde, Dresden
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Regensburg-Klinik und Poliklinik für Augenheilkunde, Regensburg
  - Universitäts-Augenklinik Tübingen, Tübingen
- India (12):
  - L V Prasad Eye Institute, Hyderabad, Andhra Pradesh
  - L V Prasad Eye Institute, Visakhapatnam, Andhra Pradesh
  - Sri Sankaradeva Nethralaya, Guwahati, Assam
  - Narayana Nethralaya, Bangalore, Karnataka
  - PBMA'S H. V. Desai Eye Hospital, Pune, Maharashtra
  - L V Prasad Eye Institute, Bhubaneswar, Odisha
  - Sankara Nethralaya (Vision Research Foundation), Chennai, Tami Nadu
  - Aravind Eye Hospital, Madurai, Tamil Nadu
  - Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow, Uttar Pradesh
  - ICARE Research Centre and Post Graduate Institute, Noida, Uttar Pradesh
  - Dr. Rajendra Prasad Centre for Ophthalmic Sciences, A.I.I.M.S., New Delhi
  - Datta Meghe Institute of Medical Sciences, Wardha
- Israel (7):
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Soroka University Medical Center, Beersheba
  - Bnai Zion Medical Center, Haifa
  - Rabin Medical Center, Belinson Campus, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - The Tel-Aviv Sourasky Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Italy (5):
  - AOU Policlinico S. Orsola-Malpighi, Bologna
  - AOU Careggi, Florence
  - Scientific Institute Auxologico Italiano, Milan
  - Scientific institute San Raffaele, Milan
  - University Eye Clinic, Parma
- Singapore (2):
  - Singapore National Eye Centre, Singapore
  - Tan Tock Seng Hospital, Department of Ophthalmology, Singapore

REFERENCES:
- [Derived] Davis JL. The Blunt End: Surgical Challenges of Gene Therapy for Inherited Retinal Diseases. Am J Ophthalmol. 2018 Dec;196:xxv-xxix. doi: 10.1016/j.ajo.2018.08.038. Epub 2018 Sep 5. PMID 30194931